CLINICAL TRIAL: NCT01819740
Title: Analysis of a New Biomarker for Prostate Cancer Diagnosis
Acronym: HEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, MIRIAM BARRIO MUÑOZ, UROLOGY RESIDENT, Hospital de Sabadell
Other Study IDs: CSPT/URO/2013/PROSTATE
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Patients With Suspected Prostate Cancer
MeSH Terms: interventions — Seeds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients with suspected prostate cancer
  Interventions: Other: determine the levels of the "HEM" substance in seminal plasma

INTERVENTIONS:
Other: determine the levels of the "HEM" substance in seminal plasma

SUMMARY:
The aim of our study is to determine if the levels of the "HEM" substance in seminal plasma are associated with the presence of prostate cancer in transrectal prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or laboratory suspected of prostate cancer

Exclusion Criteria:

* Inability to ejaculate

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with clinical or laboratory suspected of prostate cancer attends in Parc Tauli Universitary Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
substance "HEM" concentration in seminal plasma (mEq/L measured by spectro-photometry | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Barrio-Muñoz, Principal Investigator — Hospital Universitario Parc Tauli de Sabadell. Spain
Locations (1):
- Hospital Universitario Parc Taulí, Sabadell, Barcelona, Spain